CLINICAL TRIAL: NCT04016285
Title: Comparison to Short-duration Tourniquet Total Knee Arthroplasty (TKA) With the Aquamantys® Bipolar Sealer and the Standard of Care in the Setting of Outpatient TKA: A Randomized, Double-blinded Study
Brief Title: Total Knee Replacement With Tourniquet or Aquamantys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Duncan (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Stephen Duncan, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47988
Record Dates: First submitted 2019-06-14; First posted 2019-07-11 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Knee Replacement
Keywords: Tourniquet; Aquamantys; Arthroplasty; Total Knee; Standard of Care Tourniquet
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aquamantys (Experimental): The Aquamantys bipolar sealer is a device used during surgery to help reduce bleeding in the joint. The system uses radiofrequency energy and sterile saline (salt water) to close small blood vessels in the knee to help reduce bleeding.
  Interventions: Device: Aquamantys
- Standard of Care: Tourniquet (Active Comparator): Standard of care for reducing bleeding during the total knee arthroplasty
  Interventions: Device: Tourniquet

INTERVENTIONS:
Device: Aquamantys — The Aquamantys bipolar sealer is a device used during surgery to help reduce bleeding in the joint. The system uses radiofrequency energy and sterile saline (salt water) to close small blood vessels in the knee to help reduce bleeding.
  Arms: Aquamantys
Device: Tourniquet — Standard of care for reducing bleeding during the total knee arthroplasty
  Arms: Standard of Care: Tourniquet

SUMMARY:
The purpose of this study is to compare quadriceps muscle strength, pain, opioid consumption and patient function during the first three months after short-stay total knee replacement between patients treated with short-duration tourniquet knee replacement with the Aquamantys® bipolar sealer versus those treated with the standard of care (tourniquet used throughout the case and no Aquamantys®).

By doing this study, investigators hope to learn if short duration tourniquet knee replacement with the Aquamantys® bipolar sealer is more effective than standard of care (tourniquet used throughout the case and no Aquamantys®). The purpose of this study is to compare quadriceps muscle strength, pain, opioid consumption and patient function during the first three months after short-stay total knee replacement between patients treated with short-duration tourniquet knee replacement with the Aquamantys® bipolar sealer versus those treated with the standard of care (tourniquet used throughout the case and no Aquamantys®).

ELIGIBILITY:
Inclusion Criteria:

* primary total knee arthroplasty

Exclusion Criteria:

* repeat knee replacement (revision arthroplasty)
* bilateral knee replacements on the same day
* partial knee replacements
* health or social limitations that do not allow for the participant to be discharged to home on the same day or day after surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Duncan, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentcuky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
We do not have permission to share the IPD

REFERENCES:
- [Derived] Ahmed I, Chawla A, Underwood M, Price AJ, Metcalfe A, Hutchinson C, Warwick J, Seers K, Parsons H, Wall PD. Tourniquet use for knee replacement surgery. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012874. doi: 10.1002/14651858.CD012874.pub2. PMID 33316105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients at a large, academic hospital clinic seen in the practice of an early-career, fellowship-trained arthroplasty surgeon were screened for enrollment from 2019-2022. Patients between 18 and 85 years of age being scheduled for unilateral, elective primary TKA, and competent to provide informed consent and participate in the required testing and questionnaires at follow-up appointments were invited. Patients undergoing revision TKA or unicompartmental arthroplasty were excluded.
Groups:
- Aquamantys: The Aquamantys bipolar sealer is a device used during surgery to help reduce bleeding in the joint. The system uses radiofrequency energy and sterile saline (salt water) to close small blood vessels in the knee to help reduce bleeding.
  Subjects in this arm received total knee arthroplasty with the use of the Aquamantys bipolar sealer to aid in hemostasis.
- Tourniquet: Pneumatic tourniquet use is a common practice for reducing bleeding during total knee arthroplasty
  Subjects in this arm received total knee arthroplasty with the use of a pneumatic tourniquet to aid in hemostasis.
Period: Overall Study
Arm/Group | Aquamantys | Tourniquet
Started | 36 | 37
Completed | 29 | 29
Not Completed | 7 | 8
Not completed — Did not progress to surgery | 2 | 5
Not completed — Failed to collect outcome data | 5 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population differs from the total enrollment of 73 because seven participants initially consented for surgery ultimately did not progress to that point.
  Additionally, this number is greater than the 58 documented as completing the study. This was due to high turnover in research staff during the COVID-19 pandemic, which resulted in no outcome data being collected for eight participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aquamantys | Tourniquet | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Customized [Count of Participants; unit: Participants]
  44-54 years | 4 | 7 | 11
  55-64 years | 17 | 13 | 30
  65-74 years | 9 | 9 | 18
  75+ years | 4 | 3 | 7
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 13 | 15 | 28
  Woman | 21 | 17 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 25 | 30 | 55
  Black, Non-Hispanic | 5 | 1 | 6
  Asian | 1 | 0 | 1
  Hispanic | 0 | 1 | 1
  Other | 3 | 0 | 3
Body Mass Index, Categorical [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 1 | 0 | 1
  18.5-24.9 kg/m^2 | 3 | 2 | 5
  25-29.9 kg/m^2 | 17 | 18 | 35
  30-39.9 kg/m^2 | 6 | 5 | 11
  40+ kg/m^2 | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Isometric Quadriceps Strength
Description: The participant will sit in a seated position and a stabilizing strap will be placed around the bottom of the participant's shank and attached to a hand-held dynamometer. The participant will be asked to slowly kick the foot as hard as they can into the dynamometer pad (muscle testing hardware), and force will be measured. Increased measured force indicates greater quadriceps strength. Measurements will be recorded for both the operative extremity and the non-operative extremity, and the results will be expressed as a percentage of the mean strength measured in operative extremities compared to that measured in non-operative extremities for each study group.
Time Frame: 2 weeks
Population: The numbers of participants listed in this section do not match the overall number of participants listed as completing the study. This is due to lapses in data collection procedures that were brought on by high rates of research staff turnover during the COVID-19 pandemic. The numbers here reflect the number of participants in each group for whom isometric quadriceps strength was collected at two weeks in both the operative extremity and the non-operative extremity.
Measure: Mean (Standard Deviation); unit: Nm/kg
Units Other Than Participants: Lower Extremities
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 14 | 13
Number analyzed (Lower Extremities) | 28 | 26
Nm/kg | 11.58 (7.87) | 9.60 (3.33)

2. Secondary Outcome: Pain (VAS)
Description: Pain will be measured using the visual analog scale (VAS), which assess pain levels on a scale from 0-10. Lower numbers indicate less pain while higher numbers indicate more pain.
Time Frame: Preoperative, 2 weeks, 6 weeks, 12 weeks
Population: The difficulty encountered in retaining research staff, in addition to the constraints associated with the COVID-19 pandemic, led to inability to collect this data point.
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Knee Osteoarthritis (KOOS,JR)
Description: Knee injury Osteoarthritis Outcome Score, Joint Replacement (KOOS,JR) patient-reported outcome score. The KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR scores are reported here in a range from 0-28 with mean and standard deviation for each group at two and six weeks post-op. Higher scores represent better perceived knee function.
Time Frame: 2 weeks post-op, 6 weeks post-op
Population: This number differs from that listed in the primary outcome as this was a passive, participant driven outcome measure as opposed to our primary outcome, which required the presence of research staff at clinic follow up.
  It was our original intention to collect this information at 12 weeks following surgery. However, the increased pressure to reduce in-person visits during the COVID-19 pandemic necessitated a temporary change in practice and made collecting this data at 12 weeks unfeasible.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 26 | 28
Score on a scale
  Two Week KOOS, JR Score | 13 (2.2) | 10 (1.4)
  Six Week KOOS, JR Score | 16 (2.1) | 17 (1.8)

4. Secondary Outcome: Emotional Health (VR-12 MCS)
Description: The Veterans Rand-12 Mental Component Score will be used to quantify the impact of the participants emotional health on their daily activities. The VR-12 consists of 12 questions, is scored from 0-100 with lower scores indicating that emotional health has a more dramatic impact on the participant's daily life.
Time Frame: Preoperative
Population: as for outcome 2
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Knee Function Questionnaire
Description: The knee function questionnaire is a study-specific questionnaire to assess knee problems that may affect everyday life. It consists of three questions: one about walking support, one about going up stairs and one about coming down stairs. Responses are categorical, and will be used to compare the proportion of patients in each group that can walk without a walker or cane, or navigate stairs without the use of upper body support. The knee function questionnaire is not a graded scale, but will be used to assess the proportion of each group that self-reports the ability to perform these 3 tasks at each of the study time points.
Time Frame: Preoperative, 2 weeks, 6 weeks, 12 weeks
Population: as for outcome 2
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Sit to Stand Test
Description: This is a timed test used to measure mobility and function. Participants are positioned in a standard 16" office chair with their arms at their sides and back located against the back of the chair. Participants are instructed to stand and sit as quickly as possible 5 times. The test is timed using a stopwatch and the timer is stopped when the individual achieves a standing position on the 5th trial. Shorter times indicate better mobility and function.
Time Frame: 6 weeks, 12 weeks
Population: as for outcome 2
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Opioid Use
Description: Opioid use will be assessed with a single question with a binary response (either yes the participant is taking opioid medications or no they are not).
Time Frame: Preoperative, 2 weeks, 6 weeks, 12 weeks
Population: as for outcome 2
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Isometric Quadriceps Strength
Description: Strength will be assessed at multiple time points during the study. The participant will sit in a seated position and a stabilizing strap will be placed around the bottom of the participant's shank and attached to a hand-held dynamometer. The participant will be asked to slowly kick the foot as hard as they can into the dynamometer pad (muscle testing hardware) placed on the anterior aspect of the participant's distal tibia. One practice trial followed by 3 actual trials will be performed. The participant will receive a 30-second rest in between each trial and a 1-minute rest in between legs for each test to prevent fatigue. Increased measured force indicates greater quadriceps strength.
Time Frame: 6 weeks and 12 weeks
Population: as for outcome 2
Arm/Group | Aquamantys | Tourniquet
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events from the time of surgery for a total of 12 weeks.
Arm/Group | Aquamantys | Tourniquet
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32

LIMITATIONS AND CAVEATS:
Limitations encountered in this study include loss to follow up prior to subjects undergoing surgery, impacts to clinical workflow stemming from the COVID-19 pandemic, high staff turnover and subsequent impacts on data collection procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT04016285/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT04016285/ICF_001.pdf